CLINICAL TRIAL: NCT04964700
Title: Analysis of Multiple Sclerosis Patients Who Have Had Greater Than 60 Infusions of Natalizumab: Safety and Efficacy
Brief Title: Analysis of MS Patients Who Have Had Greater Than 60 Infusions of Natalizumab
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Multiple Sclerosis Center of Northeastern New York (Other)
Responsible Party: Principal Investigator, Keith Edwards, M.D., Principal Investigator, Multiple Sclerosis Center of Northeastern New York
Other Study IDs: US-TYS-11750
Record Dates: First submitted 2021-05-27; First posted 2021-07-16 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Multiple Sclerosis
Keywords: Natalizumab; Tysabri
MeSH Terms: conditions — Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Natalizumab — Monthly Infusions
  Other Names: Tysabri

SUMMARY:
The purpose of this study is to explore the safety and efficacy data in clinic patients who have been treated with Natalizumab for more than 60 continuous infusions.

DETAILED DESCRIPTION:
This is a retrospective chart review and data analysis of patients at the MS Center of Northeastern New York , P.C., who have had greater than 60 continuous infusions prior to the IRB approval date. Only records that are in existence at the time of the IRB review and approval will be accessed for inclusion in the data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis patients treated with long term use of natalizumab--60 or more infusions (5 years)

Exclusion Criteria:

* Patients who do not have 60 or more infusions (5 years) of Natalizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have received 60 or more infusions in the MS Center of Northeastern New York, P.C. Clinic will be included for analysis.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of reported cases of PML ( progressive multifocal leukoencephalopathy) | While on Natalizumab (Dosing) to one year after natalizumab use (Termination Date)
  Total number of cases of PML as reported by chart review. Progressive multifocal leukoencephalopathy (PML) is a disease of the white matter of the brain, caused by a virus infection that targets cells that make myelin--the material that insulates nerve cells (neurons).
Number of documented exacerbations | While on Natalizumab (Dosing) to one year after natalizumab use (Termination Date)
  Total number of documented exacerbations as reported in chart review . An MS exacerbation or relapse is defined as a monophasic clinical episode with patient-reported symptoms and objective findings typical of MS, reflecting a focal or multifocal inflammatory demyelinating event in the central nervous system, developing acutely or sub-acutely, with a duration of at least 24 hours, with or without recovery, and in the absence of fever or infection.
Change in EDSS Score | One year prior to natalizumab use (Baseline), while on Natalizumab (Dosing), to one year after natalizumab use (Termination Date)
  Expanded Disability Assessment- (EDSS) The EDSS is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. The scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability.
Number of new MRI lesions | While on Natalizumab (Dosing) to one year after natalizumab use (Termination Date)
  Total number of new lesions as reported on MRI (Magnetic Resonance Imaging) MRI can indicate MS disease activity by showing a pattern consistent with inflammation of active demyelinating lesions. It can show types of lesions that are new or getting bigger due to demyelination (damage to the myelin that covers certain nerves).

SECONDARY OUTCOMES:
Change in JCV Ab index value | One year prior to natalizumab use (Baseline), while on Natalizumab (Dosing), to one year after natalizumab use (Termination Date)
  Change in semi-annual JCV Ab (John Cunningham Virus Antibody) index value. The JC Virus (JCV) is associated with a increased risk of progressive multifocal leukoencephalopathy (PML). Detection of antibodies to JCV in serum or plasma is a reliable indicator of exposure to JCV.
Number of reported clinically significant changes on MRI that may indicate other opportunistic infections. | One year prior to natalizumab use (Baseline), while on Natalizumab (Dosing), to one year after natalizumab use (Termination Date)
  Number of reported clinically significant changes on MRI as reported. Magnetic Resonance Imaging (MRI) is a non-invasive imaging technology that produces three dimensional detailed anatomical images. It is often used for disease detection, diagnosis, and treatment monitoring.
Number of clinically significant lab values as measured CMP ( Comprehensive Metabolic Panel) | While on Natalizumab (Dosing), to one year after natalizumab use (Termination Date)
  A comprehensive metabolic panel (CMP) is a test that measures 14 different substances in your blood. It provides important information about your body's chemical balance and metabolism. Clinically significant changes in values will be recorded.
Number of clinically significant lab values as measured by the CBC (Complete Blood Count) | While on Natalizumab (Dosing), to one year after natalizumab use (Termination Date)
  The complete blood count (CBC) is a group of tests that evaluate the cells that circulate in blood, including red blood cells (RBCs), white blood cells (WBCs), and platelets (PLTs). The CBC can evaluate your overall health and detect a variety of diseases and conditions, such as infections, anemia and leukemia. Clinically significant changes in values will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Keith R Edwards, M.D., Principal Investigator — MS Center of Northeastern New York, P.C.
Locations (1):
- Multiple Sclerosis Center of Northeastern New York, P.C., Latham, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gunnarsson M, Malmestrom C, Axelsson M, Sundstrom P, Dahle C, Vrethem M, Olsson T, Piehl F, Norgren N, Rosengren L, Svenningsson A, Lycke J. Axonal damage in relapsing multiple sclerosis is markedly reduced by natalizumab. Ann Neurol. 2011 Jan;69(1):83-9. doi: 10.1002/ana.22247. Epub 2010 Dec 8. PMID 21280078
- [Background] Miravalle A, Jensen R, Kinkel RP. Immune reconstitution inflammatory syndrome in patients with multiple sclerosis following cessation of natalizumab therapy. Arch Neurol. 2011 Feb;68(2):186-91. doi: 10.1001/archneurol.2010.257. Epub 2010 Oct 11. PMID 20937940